CLINICAL TRIAL: NCT02720146
Title: The Effect of Platelet Lysate on Corneal Epithelial Wound healing---the Collection of Human Serum From Volunteers
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201510123RINB
Record Dates: First submitted 2016-03-21; First posted 2016-03-25 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Comparison of Epitheliotrophic Ability Between Human Serum and Commercialized Human Platelet- Cell and Animal Model
Keywords: Dry eye
MeSH Terms: conditions — Disease Models, Animal; Dry Eye Syndromes

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Artificital tear: The epitheliotrophic ability in cell and animal model
- Human peripheral serum: The epitheliotrophic ability in cell and animal model
- Human platelet lysate: The epitheliotrophic ability in cell and animal model

SUMMARY:
"Poor corneal epithelialization problem" can be found in a lot of ocular surface disorders, including limbal insufficiency, dry eye, chemical burn and neurotrophic disorders. Delayed corneal epithelialization under any circumstances can lead to corneal infection, corneal melting, corneal opacity, pain or blurred vision. It is thus important to develop pharmacological methods to promote corneal epithelial wound healing in those patients. Previously, various epitheliotrophic growth factors, autologous serum, cord blood serum, etc. have been proved to be effective in promoting corneal epithelial wound healing. However, those topical agents have the drawbacks including the difficulties during preparation, expensive price, non-standardized quality and the risk of contamination during preparation. It will be clinically important to find other blood derivatives which are effective, convenient for use, stable in quality and being cheap.

During the recent few years, various" platelet related blood derivatives" have been proved to contain a lot of epitheliotrophic growth factors, and can promote wound healing. Among those products, "platelet lysate" has the benefits of being commercially available. It can avoid the complicated producing procedure, and has stable quality. Although platelet lysate has been widely used in various medical fields, especially in culturing mesenchymal stem cells, its potential in promoting corneal epithelial wound healing has not been proven. The purpose of this project is to explore the possibility of using platelet lysate to treat patients with poor corneal epithelialization problem, and compare its epitheliotrophic ability with other blood derivatives. The cultured human corneal epithelial cell line will be used for all experiments, and will be cultured with media containing different blood products: (1) control group without blood derivatives, (2) fetal bovine serum, (3) human serum, (4) platelet lysate commercial product-UltraGro, (5)platelet lysate commercial product---PlatMax. MTS assay will be used to measure proliferation ability. "Scratch-induced directional wounding assay" and "Boyden chamber chemotaxis assa" will be used to measure cell migration. Scanning electron microscopy, transmission electron microscopy, transepithelial electric resistance (TEER) and immunohistochemistry with junctional proteins will be used to measure cellular differentiation. Through these experiments, the investigator aim to understand whether platelet lysate can replace other blood derivatives, and be used for treating patients with corneal epithelialization problem.

Beside, current medications in dry eye are all manufactured, transported and used in the form of liquid form. However, it is more disturbing in transporting, commercializing, storing and the limitation of expiration date for current medications compared with powder form medications. Therefore, improving the convenience of utilizing and storage without at the expense of the efficacy of blood-derivatives has become a critical issue. Our study also aimed at trying to produce platelet-related derivatives (including platelet lysate) and human serum into the form of dry powder and resuspended it with preservative-free artificial tears. The investigator would compare the epitheliotrophic ability of the liquid form of blood derivatives and the powder form of blood derivatives.

Since human serum is needed for comparison , the investigator proposed this IRB to collect human serum from healthy volunteers。

ELIGIBILITY:
* Healthy volunteer control without ocular surface disease or prior ophthalmic surgery history
* Healthy volunteer without any other systemic disease taking longterm medication

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Acquired whole blood for human serum used for wound healing array
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
The purpose of this project is to collect the human serum as a control group, | 1 year
  The purpose of this project is to collect the human serum as a control group, and to explore the possibility of using "platelet lysate" to treat patients with poor corneal epithelialization problem, and compare its epitheliotrophic ability with other blood derivatives. Besides, the investigator would also compared the efficacy of dry powder of platelet lysate and other blood derivatives.
  The cultured human corneal epithelial cell line will be used for all experiments, and will be cultured with media containing different blood products:
  1. control group without blood derivatives,
  2. fetal bovine serum,
  3. human peripheral blood serum
  4. platelet lysate commercial product-UltraGro
  5. platelet lysate commercial product---PlatMax.
  6. the dry powder of human peripheral blood serum resuspended with artificial tear The investigator will evaluate the effects of these blood derivatives.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Li Chen, Principal Investigator — National Taiwan University, Ophthalmologic Department
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan